CLINICAL TRIAL: NCT03940430
Title: Lactoferrin Versus Ferrous Sulfate in Management of Iron Deficiency Anemia Among Female Medical Ain Shams Students
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: yasmin gamal el gendy (Other)
Responsible Party: Sponsor-Investigator, yasmin gamal el gendy, Yasmin gamel elgendy clinical professor, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ain shams
Record Dates: First submitted 2019-04-12; First posted 2019-05-07 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; ferrous sulfate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lactoferrin in iron deficiency anemia (Active Comparator): lactoferrin ( pravotin) 100mg twice daily
  Interventions: Drug: Lactoferrin
- Ferrous sulfate in iron deficiency anemia (Active Comparator): ferrous sulphate (hemojet)
  Interventions: Drug: Ferrous sulfate
- Lactoferrin and ferrous sulfate in iron deficiency anemia (Active Comparator): Lactoferrin 100 mg twice daily and ferrous sulfate
  Interventions: Drug: Lactoferrin; Drug: Ferrous sulfate

INTERVENTIONS:
Drug: Lactoferrin — This study aims to compare the efficacy of lactoferrin versus iron supplementation versus two combined supplementation on iron deficiency anemia in female medical Ain Shams students by using iron profile.
  Arms: Lactoferrin and ferrous sulfate in iron deficiency anemia; Lactoferrin in iron deficiency anemia
Drug: Ferrous sulfate — This study aims to compare the efficacy of lactoferrin versus iron supplementation versus two combined supplementation on iron deficiency anemia in female medical Ain Shams students by using iron profile.
  Other Names: ferrous sulphate
  Arms: Ferrous sulfate in iron deficiency anemia; Lactoferrin and ferrous sulfate in iron deficiency anemia

SUMMARY:
This study aims to compare the efficacy of lactoferrin versus iron supplementation versus two combined supplementation on iron deficiency anemia in female medical Ain Shams students by using iron profile.

DETAILED DESCRIPTION:
Iron, an essential element for cell growth and proliferation, is a component of fundamental processes such as DNA replication and energy production. However, iron can also be toxic when present in excess for its capacity to donate electrons to oxygen, thus causing the generation of reactive oxygen species (ROS), such as superoxide anions and hydroxyl radicals

Prevalence of iron deficiency anemia is roughly 38% of pregnant women, 29% of non-pregnant women and 29% of all women of reproductive age have anemia globally

Human lactoferrin (hLf), an 80-kDa multifunctional iron-binding cationic glycoprotein, is constitutively secreted by exocrine glands and by neutrophils during inflammation. hLf is recognized as a key element in the host immune defense system

Bovine Lf (bLf), which shares high sequence homology with the human protein, is also a multifunctional glycoprotein with identical antibacterial, antifungal, antiviral, antiparasitic, anti-inflammatory, and immunomodulatory activities of hLf Lactoferrin is synthesized by exocrine glands and neutrophils under conditions of inflammation and at site of infection through its iron binding and formation of reactive oxygen species physiological transport of iron from tissue to circulation, thus curing iron deficiency and iron deficiency anemia

A study done for pregnant women showed an increase of total serum iron in all bovin lactoferrin treated women.

Therefore, the investigators speculated that bLf efficacy in curing AI was presumably not linked to direct iron supplementation, but to a more complex mechanism involving this protein in iron homeostasis

Lactoferrin was also proven useful for prevention of iron deficiency anemia special among female long distance runner

Lactoferrin was more effective than ferrous sulphate over a two months period in pregnant women with iron deficient anemia Aim of the Work

This study aims to compare the efficacy of lactoferrin versus iron supplementation versus two combined supplementation on iron deficiency anemia in female medical Ain Shams students by using iron profile.

ELIGIBILITY:
Inclusion Criteria:

* female student with iron deficiency anemia

Exclusion Criteria:

* clinical diagnosis of chronic disease as DM, Malabsorption disease Celiac, blood disease as thalassemia, or haemoglobinopathy

Intervention:

Study participants will be divided into 3 groups; Group 1: 35 participants will be supplemented with iron salt 324 mg (66 mg of elemental iron) orally three time per day before meal for one month Group 2: 35 participants will be supplemented with LF sachet 100 mg twice per day before meal for period of one month.

Group 3: 35 participants will be supplemented with combined iron salt 324 mg (66 mg of elemental iron) orally three time per day before meal for one month, and LF sachet 100 mg twice per day before meal for period of one month.

Ages: 19 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Management of iron deficiency anemia incidence by using lab measures include iron profile | One month
  Management of iron deficiency anemia

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin G Elgendy, M.d, Principal Investigator — Ainshams university
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No